CLINICAL TRIAL: NCT05156918
Title: The Effects of High-Intensity Exercise on Biological Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Gurinder Bains, Associate Professor School of Allied Health, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 5210437
Record Dates: First submitted 2021-11-29; First posted 2021-12-14 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Experimental): Exercise group participants will perform supervised high intensity exercise three times per week at the LLU department of physical therapy laboratory utilizing treadmills, stationary bicycles, and rowing machines.
  Interventions: Other: Exercise
- Control Group (Active Comparator): Control group participants will make no modifications to regular diet or exercise habits for 30 days.
  Interventions: Other: Non Exercise

INTERVENTIONS:
Other: Exercise — Participants will rotate between three exercise machines (randomly assigned rotation order at outset): A Concept C2 rowing machine, a stationary bicycle, and a treadmill. Study participants will use a different machine each day so that they are using each of the three exercise machines once per week. Two treadmills, two bikes, and two rowers are available during each exercise session. Participants will be randomly assigned to one of three machine orders: treadmill-rower-bike, rower-bike-treadmill, or bike-treadmill-rower. We will employ a percent of heart rate protocol as an exercise intensity measure (77-93% of age-adjusted maximum heart rate) rather than a less well-defined maximal effort protocol or rating of perceived exertion scale. For the purposes of this exercise protocol high intensity exercise will be defined as 77-93% of age adjusted maximum heart rate.
  Arms: Exercise Group
Other: Non Exercise — There are no modifications to regular diet or exercise habits for 30 days.
  Arms: Control Group

SUMMARY:
The purpose of this graduate student research study is to determine if a high-intensity exercise program can slow or reverse biological (transcriptomic) aging and shed light on the underlying transcriptomic pathways involved.

DETAILED DESCRIPTION:
24 males and 24 females will be randomly assigned to either the control group or the exercise group. Baseline measures will be obtained, including questionnaires (on stress, sleep, depression, activity level, and fitness), body composition measures, vital signs, and a blood draw. Control group participants will make no modifications to regular diet or exercise habits for 30 days. Exercise group participants will perform supervised high intensity exercise three times per week at the LLU department of physical therapy laboratory utilizing treadmills, stationary bicycles, and rowing machines. Results will be collected following conclusion of the 30-day study protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Sex: Both Males and Females
2. Age: 40-65 years old
3. Physical Fitness: Below average scores on the Self report fitness questionnaire
4. Physical Activity: Low as measured by the International Physical Activity Questionnaire

Exclusion Criteria:

1. Prior (within the last 5 years) or current history of cardiovascular disease, stroke, unexplained weight loss, clinical depression, congestive heart failure, cancer, arrythmia, respiratory disease, or other serious medical conditions that would make exercise unsafe or prevent full participation in the exercise protocol.
2. Any self-reported significant increase or decrease in activity levels within the past thirty days.
3. Current use of the following medications: antibiotics, glucocorticoids, anticoagulants, narcotics, antiepileptic medications, antipsychotics, antidepressants, and hypoglycemic agents.
4. Current self-reported pregnancy

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-06-28 (Actual)

PRIMARY OUTCOMES:
venipuncture procedure | Change between baseline and 30 days
  Participants will have 8ml of blood drawn on two separate occasions by a certified phlebotomist. The first 8 ml (1.62tsp) blood draw will occur at 8am on day 1 of the study protocol. The second 8ml (1.62tsp) blood draw will occur approximately 30 days later. The total blood draw volume will be 16ml or approximately 3.25 teaspoons. The blood draw is to test for the effects of exercise on gene expression and aging.

SECONDARY OUTCOMES:
Perceived stress scale survey | Change between baseline and 30 days
  The most widely used psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are regarded as stressful during the past 30 days. Responses are scored from 0 to 4. And the total score can be from 0 to 40.
  "Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress."
Pittsburgh Sleep Quality Index | Change between baseline and 30 days
  A self-rated questionnaire which assesses sleep quality over a 1-month period. Questions are scored between a zero and three. A total score of 5 or greater means poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Gurinder Bains, PhD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University, Loma Linda, California, United States